CLINICAL TRIAL: NCT02242981
Title: Disposition of [14C]-LY2623091 Following Oral Administration in Healthy Subjects
Brief Title: A Study of How the Body Breaks Down and Eliminates LY2623091
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15517; I7T-MC-RMAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2623091 (Experimental): Single oral dose of LY2623091
  Interventions: Drug: LY2623091

INTERVENTIONS:
Drug: LY2623091 — Administered orally

SUMMARY:
This type of study is called a radiolabeled study. For this study, LY2623091 (study drug) has been specially prepared to contain radiolabeled carbon [^14C]. [^14C] is a naturally occurring radioactive form of the element, carbon. This study will increase understanding about how the drug appears in the blood, urine, and stool after it is administered to healthy participants. Information about any side effects that may occur will also be collected. This study will last up to 22 days for each participant, not including screening. Screening is required within 28 days prior to enrollment

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males; as determined by physical examination, clinical laboratory tests, medical history and electrocardiograms (ECGs).
* With a body mass index of 18.5 to 32.0 kilogram per square meter (kg/m^2), inclusive.

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2623091: Single dose of 25 milligrams (mg) LY2623091 containing carbon-14 [¹⁴C]-LY2623091 (approximately 100 microcuries [µCi]) administered orally.
Period: Overall Study
Arm/Group | LY2623091
Started | 6
Received Study Drug | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants who received study drug.
Groups:
- LY2623091: Single dose of 25 mg LY2623091 containing [¹⁴C]-LY2623091 (approximately 100 µCi) administered orally.
Arm/Group | LY2623091
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Urinary and Fecal Excretion of LY2623091 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: Cumulative percent of radioactive dose recovered in urine and feces after administration at specified intervals.
Time Frame: Screening (urine only), Day -1, Day 1 (0 to 6, 6 to 12, and 12 to 24 hours), and at 24 hour intervals thereafter until the study release criteria have been met (up to 504 hours)
Population: All participants who received study drug and had quantifiable levels of radioactivity in urine and feces.
Measure: Mean (Standard Deviation); unit: percentage of radioactive dose recovered
Arm/Group | LY2623091
Number analyzed (Participants) | 6
percentage of radioactive dose recovered
  Feces | 60.5 (4.27)
  Urine | 1.39 (0.454)

2. Secondary Outcome: Plasma Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration (AUC[0-tlast]) of LY2623091
Time Frame: Day 1 (predose, 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose), 24 hours postdose, and every 24 hours thereafter until study release criteria have been met (up to 504 hours)
Population: All participants who received study drug and had evaluable AUC(0-tlast) values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | LY2623091
Number analyzed (Participants) | 6
nanograms*hour/milliliter (ng*h/mL) | 11800 (38)

3. Secondary Outcome: Plasma Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf]) of LY2623091
Time Frame: as for outcome 2
Population: All participants who received study drug and had evaluable AUC(0-inf) values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LY2623091
Number analyzed (Participants) | 6
ng*h/mL | 11800 (38)

4. Secondary Outcome: Plasma Pharmacokinetics: Maximum Concentration (Cmax) of LY2623091
Time Frame: as for outcome 2
Population: All participants who received study drug and had evaluable Cmax values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LY2623091
Number analyzed (Participants) | 6
ng/mL | 482 (15)

5. Secondary Outcome: Total Number of Metabolites of LY2623091 in Plasma, Urine, and Feces
Time Frame: Day 1 (predose, 2, 3, 4, 6, 8, and 12 hours postdose), and at 24 and 48 hours postdose
Population: All participants who received study drug and had evaluable plasma, urine, and fecal samples.
Measure: Number; unit: metabolites
Arm/Group | LY2623091
Number analyzed (Participants) | 6
metabolites
  Plasma | 7
  Urine | NA — Urine was not profiled due to the low percentage of dose excreted in urine.
  Feces | 17

ADVERSE EVENTS:
Description: Includes serious adverse events (SAEs) and all other non-serious adverse events (AEs) that met the frequency threshold regardless of causality.
Arm/Group | LY2623091
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2623091 (N=6)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days